CLINICAL TRIAL: NCT06953856
Title: Effect of Occlusal Reduction on Post-operative Pain of Symptomatic and Asymptomatic Molar Teeth
Brief Title: Analyzing the Impact of Occlusal Reduction on the Pain Following Root Canal Therapy in Molar Teeth With and Without Pain in Turkish Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, AYSENUR KAMACI ESEN, Assistant Professor, Sakarya University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: E-71522473-050.01.04-39802-329
Record Dates: First submitted 2025-04-05; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Irriversible Pulpitis
Keywords: Analgesics; Occlusal reduction; Postoperative pain; Single-visit endodontic treatment
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Occlusal reduction, (Other): one of the group received occlusal reduction after root canal treatment while other did not.
  Interventions: Other: occlusal reduction
- no occlusal reduction (No Intervention): this group did not receive any occlusal reduction after root canal treatment.

INTERVENTIONS:
Other: occlusal reduction — Occlusal reduction is a procedure that applied patients for different aims. One of these aims is pain relief after endodontic treatment and there are some studies about this topic however, there is no consensus about it. This discrepency could be related to differences of the inclusion criteria for this reason this study aimed to get a reliable result.
  Other Names: occlusal reduction procedure
  Arms: Occlusal reduction,

SUMMARY:
Introduction: This study aimed to compare the intensity of postoperative pain after single-visit root canal treatment of symptomatic or asymptomatic teeth following occlusal reduction.

Methods: A total of 140 symptomatic or asymptomatic patients in need of root canal therapy were registered in this prospective, single-center, single-blind, randomized clinical trial.

For all patients, root canal treatment was carried out in a single visit, and the teeth were restored using composite resin. The teeth were randomly allocated into two equal groups according to whether occlusal reduction was done or not. The patients' pain were assessed using a 0-3 verbal rate scale 1, 3, and 7 days following root canal treatment. The pain incidence and intensity were compared using the chi-square and Fisher's exact tests.

DETAILED DESCRIPTION:
Root canal treatments is usually associated with post-operative pain and this is a bothersome situation for both patient and practitioner. Due to this reason number of researches focus on the factors that may relief patients pain. Occlusal reduction is one of the factors that means the chewing surface of the teeth are cut off and no longer in contact.Despite the large number of studies on this subject, no consensus has been reached. Decoupling group standardization and arriving at a more consistent conclusion were the goals of this research. The aim of this research is to evaluate the impact of occlusal reduction on postoperative pain in both symptomatic and asymptomatic molar teeth.

ELIGIBILITY:
Inclusion Criteria:

* Healty patients
* Maxillary and mandibulary first and second molars
* Irriversible pulpitis cases with or without prior discomfort

Exclusion Criteria:

* Patients under 18 years old,
* Patients older 65 years old,
* Teeth with previously undergone root canal treatment,
* Complicating systemic diseases,
* Allergies o local anesthetic agents,
* Presence of acute apical apsesses,
* History of trauma,
* Analgesic, antibiotic or antiinflamatory intake 7 days before treatment,
* Periodontal pockets deeper than 4 mm,
* Multiple teeth that require endodontic treatment,
* Pregnancy,
* Teeth that can not be restored,
* Patients who needed emergency treatment,
* Grade 2 or 3 mobility,
* Patients with bruxism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Effect of occlusal reduction on pain relief | from enrollment to the end each patient called for a week to understand their pain levels and each of them called after 1st, 3th, 7th days treatment.
  This study was primarily aim to understand the effect of occlusal reduction on pain relief after root canal treatment of irriversible pulpitis. After root canal treatment patients were called to estimate their pain levels. A 0-3 rate verbal rating scale was used for this aim.
  0: no discomfort or pain
  1. mild pain (not requiring analgesic medication)
  2. moderate pain (requiring analgesic medication)
  3. severe pain (interfering with physical activity and minimally responsive to analgesics)

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University Facultry of Dentistry, Adapazarı, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Parirokh M, Rekabi AR, Ashouri R, Nakhaee N, Abbott PV, Gorjestani H. Effect of occlusal reduction on postoperative pain in teeth with irreversible pulpitis and mild tenderness to percussion. J Endod. 2013 Jan;39(1):1-5. doi: 10.1016/j.joen.2012.08.008. Epub 2012 Sep 29. PMID 23228248
- [Background] Ahmed YE, Emara RS, Sarhan SM, El Boghdadi RM, El-Bayoumi MAA, El-Far HMM, Sabet NE, Abou El-Nasr HM, Gawdat SI, Amin SAW. Post-treatment endodontic pain following occlusal reduction in mandibular posterior teeth with symptomatic irreversible pulpitis and sensitivity to percussion: a single-centre randomized controlled trial. Int Endod J. 2020 Sep;53(9):1170-1180. doi: 10.1111/iej.13328. Epub 2020 Jun 15. PMID 32418236
- [Background] Emara RS, Abou El Nasr HM, El Boghdadi RM. Evaluation of postoperative pain intensity following occlusal reduction in teeth associated with symptomatic irreversible pulpitis and symptomatic apical periodontitis: a randomized clinical study. Int Endod J. 2019 Mar;52(3):288-296. doi: 10.1111/iej.13012. Epub 2018 Sep 28. PMID 30171777
- [Background] Rosenberg PA, Babick PJ, Schertzer L, Leung A. The effect of occlusal reduction on pain after endodontic instrumentation. J Endod. 1998 Jul;24(7):492-6. doi: 10.1016/S0099-2399(98)80054-X. PMID 9693578
- [Background] Nguyen-Nhon D, Nagendrababu V, Pulikkotil SJ, Rossi-Fedele G. Effect of occlusal reduction on postendodontic pain: A systematic review and meta-analysis of randomised clinical trials. Aust Endod J. 2020 Aug;46(2):282-294. doi: 10.1111/aej.12380. Epub 2019 Oct 22. PMID 31638301
- [Background] Sathorn C, Parashos P, Messer H. The prevalence of postoperative pain and flare-up in single- and multiple-visit endodontic treatment: a systematic review. Int Endod J. 2008 Feb;41(2):91-9. doi: 10.1111/j.1365-2591.2007.01316.x. Epub 2007 Oct 23. PMID 17956561